CLINICAL TRIAL: NCT02054156
Title: OPTIMIZing Treatment for Early Pseudomonas Aeruginosa Infection in Cystic Fibrosis: The OPTIMIZE Multicenter, Placebo-Controlled, Double-Blind, Randomized Trial
Brief Title: OPTIMIZing Treatment for Early Pseudomonas Aeruginosa Infection in Cystic Fibrosis
Acronym: OPTIMIZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bonnie Ramsey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Bonnie Ramsey, Professor of Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPTIMIZE-IP-12; 1U01HL114623-01A1 (NIH); 1U01HL114589-01A1 (NIH)
Record Dates: First submitted 2014-02-01; First posted 2014-02-04 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis (CF); Azithromycin; Tobramycin solution for inhalation (TIS); Pseudomonas aeruginosa (Pa); Early Pseudomonas aeruginosa infection; Pulmonary exacerbation; Standardized anti-pseudomonal therapy
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Azithromycin; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azithromycin and TIS (Active Comparator): azithromycin and tobramycin solution for inhalation (TIS) Azithromycin 3 times weekly, oral suspension, 10 mg/kg/dose up to 500 mg, for 18 months Tobramycin solution for inhalation (TIS), 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
  Interventions: Drug: azithromycin; Drug: Tobramycin solution for inhalation
- placebo and TIS (Placebo Comparator): placebo and tobramycin solution for inhalation (TIS) Placebo 3 times weekly, oral suspension, volume-matched to azithromycin, for 18 months Tobramycin solution for inhalation (TIS), 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
  Interventions: Drug: placebo; Drug: Tobramycin solution for inhalation

INTERVENTIONS:
Drug: azithromycin — 3 times weekly, oral suspension, 10 mg/kg/dose up to 500 mg, for 18 months
  Arms: azithromycin and TIS
Drug: placebo — 3 times weekly, oral suspension, volume-matched to azithromycin, for 18 months
  Arms: placebo and TIS
Drug: Tobramycin solution for inhalation — 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
  Other Names: TIS

SUMMARY:
The purpose of this trial is to compare the effects of treatment with tobramycin solution for inhalation (TIS) with and without azithromycin in people with cystic fibrosis (CF) age 6 months to 18 years who have early isolation of Pseudomonas aeruginosa (Pa) from a respiratory culture. Specimens of blood and sputum or throat swabs will be taken during the study along with pulmonary function testing. Participants will receive initial treatment with TIS followed additional treatment with TIS if quarterly respiratory cultures are positive for Pa in addition to either azithromycin or placebo for 18 months.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) lung disease begins in the first few months of life and follows a course of recurrent lower airway bacterial infection and inflammation and progression of disease over years and decades at a variable pace. With the development of chronic lung infection, obstructive disease progressively worsens, ultimately leading to respiratory failure. Pseudomonas aeruginosa (Pa) is the most important pathogen infecting the CF lower airways, and its acquisition early in life is associated with a pro-inflammatory effect, lower lung function, poor nutritional outcomes, and decreased survival.

Pseudomonas aeruginosa (Pa) infection of the cystic fibrosis (CF) airway typically proceeds from early infection to chronic infection. Although some studies have shown that a minority of individuals with CF spontaneously clear early Pseudomonas aeruginosa (Pa) infection, data from multiple studies suggest that antibiotics are superior to no treatment in clearing Pseudomonas aeruginosa (Pa) from respiratory cultures. Understanding the transition period from early to chronic Pseudomonas aeruginosa (Pa) infection is thus of critical importance in identifying strategies to prevent this progression.

The study will assess the clinical and microbiologic efficacy and safety of azithromycin given three times weekly in combination with standardized tobramycin solution for inhalation (TIS) therapy among children with early Pseudomonas aeruginosa (Pa). TIS therapy is defined as an initial eradication treatment with 1-2 courses of 28 days TIS and subsequent 28 day treatments only at times a quarterly respiratory culture is positive for Pseudomonas aeruginosa (Pa). Eligible participants will be randomized within one month of their Pseudomonas aeruginosa (Pa) positive culture to receive one of the following two treatment strategies for 18 months: (1) oral placebo in addition to standardized TIS therapy, or (2) oral azithromycin in addition to standardized TIS therapy.

At the first study visit, participants will undergo a physical examination and a review of their medical history. Lung function will be measured via spirometry (in children greater than four years of age who are able to perform spirometry), electrocardiogram (ECG) testing will be conducted, and hearing ability will be measured via audiometry. Blood will be drawn for laboratory tests and a specimen will be obtained for a respiratory culture before randomization and study drug dispensing occurs. Subsequent study visits will take place at Day 21, Weeks 13, 26, 39, 52, 65, and 78. At each visit, participants will undergo a physical examination, a spirometry test (as appropriate), a respiratory specimen for Pseudomonas aeruginosa (Pa) culture will be collected and study drug will be dispensed (except at Week 78). Participants will complete self-report or parent-completed respiratory symptom questionnaires and signs and symptoms evaluations will be performed at all visits. Repeat hearing and laboratory tests will be performed at Weeks 39 and 78 and ECG testing will be repeated at Day 21 and Week 78. Participants will be required to maintain a medication diary throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 months to ≤ 18 years
* Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype or positive CF Newborn Screening result for immunoreactive trypsinogen (IRT) IRT/DNA or IRT/IRT and one or more of the following criteria:
* sweat chloride ≥ 60 milliequivalent (mEq)/liter by quantitative by pilocarpine iontophoresis test (QPIT)
* two well-characterized mutations in the cystic fibrosis transmembrane conductive regulator (CFTR) gene
* Abnormal nasal potential difference (NPD) (change in NPD in response to a low chloride solution and isoproteronol of less than - 5 mV)
* Documented new positive oropharyngeal, sputum or lower respiratory tract culture for Pa within 30 days of the Baseline Visit (Visit 1), defined as: a) first lifetime documented Pa positive culture; or b) Pa recovered after at least a two-year history of Pa negative respiratory cultures (≥ 1 culture/ year)
* Clinically stable with no evidence of any significant respiratory symptoms at the Baseline Visit that would require administration of intravenous anti- pseudomonal antibiotics, oxygen supplementation, and/or hospitalization as determined by the study physician
* Written informed consent obtained from participant or participant's legal representative (and assent when applicable) and ability for participant to comply with the requirements of the study

Exclusion Criteria:

* Macrolide antibiotic use within 30 days of the Baseline Visit
* Initiation of current course of treatment with TIS >14 days prior to Baseline Visit
* Weight <6.0 kg at the Baseline Visit
* History of aminoglycoside hypersensitivity or adverse reaction to inhaled aminoglycoside
* History of azithromycin hypersensitivity or adverse reaction to azithromycin or allergy to macrolide antibiotics
* History of positive respiratory culture for Non-tuberculous mycobacteria (NTM) or Burkholderia cepacia complex within 2 years of the Baseline Visit
* History of unresolved, abnormal renal function (defined as serum creatinine greater than 1.5 times the upper limit of normal for age).
* History of unresolved, abnormal liver function tests (defined as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than 4 times the upper limit of normal range) or history of portal hypertension
* History of unresolved, abnormal neutropenia (ANC ≤ 1000)
* Abnormal ECG test at the Baseline Visit defined as a QT interval corrected (QTc) (B) of ≥460 msec or history of ventricular arrhythmia
* History of abnormal hearing sensitivity defined as hearing threshold levels >25 dB HL (decibels Hearing Level) for visual reinforcement audiometry (VRA) at any frequency (500-4000Hz) or >20 Decibels Hearing Level (dBHL) for play or standard audiometry at any two frequencies (500-8000Hz) in either ear, not associated with middle ear disease (including infection) or a flat (Type B) tympanogram
* New initiation of chronic therapy (greater than 21 days) with drugs known to prolong QT interval (refer to Appendix III) within 30 days prior to the Baseline Visit or coadministration of nelfinavir or oral anticoagulants
* Positive serum or urine pregnancy test at the Baseline Visit (to be performed on all females of child-bearing potential) or for females of child bearing potential: pregnant, breastfeeding, or unwilling to use barrier contraception during participation in the study
* Administration of any investigational drug within 30 days prior to the Baseline Visit
* Presence of a condition or abnormality (e.g., pre-existing heart disease) that in the opinion of the site investigator would compromise the safety of the participant or the quality of the data

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 2014-06; Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ramsey, MD, Principal Investigator — Seattle Children's Center for Clinical and Translational Research, CF Therapeutics Development Network Clinical Coordinating Center; Nicole Hamblett, PhD, Principal Investigator — Seattle Children's Core for Biomedical Statistics
Locations (45):
- United States (45):
  - CFF Affiliate Program Providence Medical Center, Anchorage, Alaska
  - CFF Care Center Arizona Health Science Center, Tucson, Arizona
  - CFF Care Center & Pediatric Program Arkansas Children's Hospital, Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - CFF Care Center & Pediatric Program Stanford University, Palo Alto, California
  - CFF Care Center & Pediatric Program Children's Hospital Colorado, Aurora, Colorado
  - CFF Care Center & Pediatric Program Yale University, New Haven, Connecticut
  - CFF Care Center & Pediatric Program Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - CFF Care Center & Pediatric Program All Children's Hospital, St. Petersburg, Florida
  - CFF Care Center & Pediatric Program Emory University, Atlanta, Georgia
  - CFF Affiliate Program Children's Healthcare of Atlanta, Atlanta, Georgia
  - CFF Care Center St. Luke's CF Clinic, Boise, Idaho
  - CFF Care Center & Pediatric Program Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - CFF Care Center & Pediatric Program Riley Hospital for Children, Indianapolis, Indiana
  - CFF Care Center & Pediatric Program University of Iowa, Iowa City, Iowa
  - CFF Care Center & Pediatric Program Maine Medical Center, Portland, Maine
  - CFF Care Center & Pediatric Program Children's Hospital Boston, Boston, Massachusetts
  - CFF Care Center & Pediatric Program University of Michigan, Ann Arbor, Michigan
  - CFF Care Center & Pediatric Program Children's Hospital of Michigan, Detroit, Michigan
  - CFF Care Center The Children's Mercy Hospital, Kansas City, Missouri
  - CFF Care Center & Pediatric Program Cardinal Glennon Children's Hospital/Saint Louis University, St Louis, Missouri
  - CFF Care Center & Pediatric Program St. Louis Children's Hospital, St Louis, Missouri
  - CFF Care Center & Pediatric Program University of Nebraska Medical Center, Omaha, Nebraska
  - CFF Care Center & Pediatric Program Monmouth Medical Center, Long Branch, New Jersey
  - CFF Care Center & Pediatric Program Columbia University, New York, New York
  - CFF Care Center & Pediatric Program SUNY Upstate Medical University, Syracuse, New York
  - CFF Care Center New York Medical College, Valhalla, New York
  - CFF Care Center & Pediatric Program University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - CFF Care Center & Pediatric Program Akron Children's Hospital, Akron, Ohio
  - CFF Care Center & Pediatric Program Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - CFF Care Center & Pediatric Program Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - CFF Care Center & Pediatric Program Nationwide Children's Hospital, Columbus, Ohio
  - CFF Care Center & Pediatric Program The Children's Medical Center, Dayton, Ohio
  - CFF Care Center & Pediatric Program Oregon Health & Sciences University, Portland, Oregon
  - CFF Care Center & Pediatric Program Hershey Medical Center, Hershey, Pennsylvania
  - CFF Care Center & Pediatric Program Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - CFF Care Center & Pediatric Program Sanford USD Medical Center, Sioux Falls, South Dakota
  - CFF Care Center & Pediatric Program University of Tennessee, Memphis, Tennessee
  - CFF Care Center & Pediatric Program Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Utah, Salt Lake City, Utah
  - CFF Care Center & Pediatric Program Children's Hospital of the King's Daughters, Norfolk, Virginia
  - CFF Care Center Medical College of Virginia, Richmond, Virginia
  - CFF Care Center & Pediatric Program Seattle Children's Hospital, Seattle, Washington
  - CFF Care Center & Pediatric Program University of Wisconsin, Madison, Wisconsin
  - CFF Care Center & Pediatric Program Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mayer-Hamblett N, Retsch-Bogart G, Kloster M, Accurso F, Rosenfeld M, Albers G, Black P, Brown P, Cairns A, Davis SD, Graff GR, Kerby GS, Orenstein D, Buckingham R, Ramsey BW; OPTIMIZE Study Group. Azithromycin for Early Pseudomonas Infection in Cystic Fibrosis. The OPTIMIZE Randomized Trial. Am J Respir Crit Care Med. 2018 Nov 1;198(9):1177-1187. doi: 10.1164/rccm.201802-0215OC. PMID 29890086

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: azithromycin and tobramycin solution for inhalation (TIS) Azithromycin 3 times weekly, oral suspension, 10 mg/kg/dose up to 500 mg, for 18 months Tobramycin solution for inhalation (TIS), 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
  azithromycin: 3 times weekly, oral suspension, 10 mg/kg/dose up to 500 mg, for 18 months
  Tobramycin solution for inhalation: 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
- Placebo: placebo and tobramycin solution for inhalation (TIS) Placebo 3 times weekly, oral suspension, volume-matched to azithromycin, for 18 months Tobramycin solution for inhalation (TIS), 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
  placebo: 3 times weekly, oral suspension, volume-matched to azithromycin, for 18 months
  Tobramycin solution for inhalation: 300 mg, twice daily for 28 days when respiratory cultures are found positive for Pa at study visits for 18 months
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 110 | 111
Completed | 35 | 30
Not Completed | 75 | 81

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.1 (5.1) | 6.8 (5.0) | 6.9 (5.0)
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution: >= 6 months - 3 years | 39 | 41 | 80
  Age Distribution: > 3 years - 6 years | 22 | 23 | 45
  Age Distribution: > 6 years - 12 years | 30 | 29 | 59
  Age Distribution: > 12 years | 19 | 18 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 104
  Male | 55 | 62 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 100 | 94 | 194
  Race: Hispanic or Latino | 5 | 10 | 15
  Race: Black or African-American | 4 | 6 | 10
  Race: Asian or Pacific Islander | 1 | 0 | 1
  Race: Unknown/Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 110 | 111 | 221
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants] — Other refers to participants with either two known, non-F508 del CF mutations, or one known, non-F508 del CF mutation and one unidentified allele which has not been classified as a CF mutation. Unidentified refers to participants with 2 alleles that have not been classified as CF mutations.
  Participants
    F508 del Homozygous | 59 | 57 | 116
    F508 del Heterozygous | 35 | 44 | 79
    Other | 11 | 9 | 20
    Unidentified | 0 | 0 | 0
    Not Available | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to a Protocol-defined Pulmonary Exacerbation
Description: Time to a protocol-defined pulmonary exacerbation requiring oral, inhaled, or intravenous antibiotics, using a prespecified definition available in the study protocol.
Time Frame: Over the 18-month study period
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 110 | 111
years | 1.350 [0.898 to NA] — Too few events occurred to estimate the upper confidence bound | 0.758 [0.572 to 0.969]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.0043, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.37 to 0.83] — The estimate is adjusted for age strata (>=6 months - 3 years, >3 - 6 years, >6 - 12 years, and >12 - 18 years)

2. Secondary Outcome: Time to Pseudomonas Aeruginosa (Pa) Recurrence
Description: Time to Pseudomonas aeruginosa (Pa) recurrence after the first quarter of treatment
Time Frame: Over the 18-month study period
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 103 | 97
years | 1.51 [0.76 to NA] — Too few events occurred to estimate the upper confidence bound | 1.46 [0.78 to NA] — Too few events occurred to estimate the upper confidence bound
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.9915, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.64 to 1.55] — The estimate is adjusted for age strata (>=6 months - 3 years, >3 - 6 years, >6 - 12 years, and >12 - 18 years)

3. Secondary Outcome: Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The number and percentage of participants with at least one event over the 18-month study period.
Time Frame: Over the 18-month study period
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 110 | 111
Participants
  Number of Participants with AE | 102 | 98
  Number of Participants with SAE | 25 | 28
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.7531, Fisher Exact; Difference in % of Participants with SAE = -2.5, 95% CI 2-sided [-13.7 to 8.7] — 95% confidence interval calculated using the Newcombe-Wilson method without continuity correction
Statistical Analysis 2: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.3593, Fisher Exact; Difference in % of Participants with AE = 4.4, 95% CI 2-sided [-3.5 to 12.6] — 95% confidence interval calculated using the Newcombe-Wilson

4. Secondary Outcome: Rate of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Rate is defined as the number of events per participant follow-up month.
Time Frame: Over the 18-month study period
Measure: Number; unit: events per participant-month
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 110 | 111
events per participant-month
  Number of AEs per participant month | 0.92 | 1.06
  Number of SAEs per participant month | 0.06 | 0.05
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Rate Ratio for Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in months. The total number of follow-up months of all participants (not per participant) in the trial was as follows: in the Azithromycin group was 1267.73 and in the Placebo group was 1193.72; Test type: Superiority; p = 0.0004, Poisson Regression; Rate Ratio = 0.86, 95% CI 2-sided [0.80 to 0.94]
Statistical Analysis 2: Comparison: Azithromycin vs Placebo; Rate Ratio for Serious Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in months. The total number of follow-up months of all participants (not per participant) in the trial was as follows: in the Azithromycin group was 1267.73 and in the Placebo group was 1193.72; Test type: Superiority; p = 0.2098, Poisson Regression; Rate Ratio = 1.25, 95% CI 2-sided [0.88 to 1.78]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/111
Serious Adverse Events (participants affected / at risk) | 25/110 | 28/111
Other Adverse Events (participants affected / at risk) | 99/110 | 92/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=110) | Placebo (N=111)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (2)
Crepitations (General disorders) | 1 (1) | 0 (0)
Decreased activity (General disorders) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 3 (3) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 7 (8)
Forced expiratory volume decreased (Investigations) | 1 (2) | 1 (1)
Fungal test positive (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Pseudomonas test positive (Investigations) | 2 (2) | 0 (0)
Pulmonary function test decreased (Investigations) | 6 (7) | 6 (6)
Respiratory syncytial virus test positive (Investigations) | 1 (1) | 0 (0)
Sputum abnormal (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=110) | Placebo (N=111)
Ear pain (Ear and labyrinth disorders) | 7 (7) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 16 (19) | 18 (21)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 13 (23)
Constipation (Gastrointestinal disorders) | 9 (13) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 16 (28) | 14 (27)
Nausea (Gastrointestinal disorders) | 4 (8) | 9 (9)
Teething (Gastrointestinal disorders) | 7 (7) | 3 (5)
Vomiting (Gastrointestinal disorders) | 27 (43) | 15 (19)
Fatigue (General disorders) | 11 (14) | 7 (8)
Pyrexia (General disorders) | 48 (94) | 35 (79)
Ear infection (Infections and infestations) | 7 (13) | 5 (7)
Otitis media (Infections and infestations) | 13 (19) | 8 (10)
Pharyngitis streptococcal (Infections and infestations) | 4 (5) | 12 (19)
Sinusitis (Infections and infestations) | 7 (10) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 14 (20) | 15 (18)
Pulmonary function test decreased (Investigations) | 6 (9) | 11 (13)
Weight decreased (Investigations) | 3 (3) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (20) | 16 (20)
Headache (Nervous system disorders) | 23 (35) | 19 (44)
Lethargy (Nervous system disorders) | 2 (2) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 70 (185) | 74 (220)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 10 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (41)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 36 (54) | 32 (71)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 15 (38)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (7)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 8 (18) | 16 (23)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 34 (81) | 36 (90)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (12)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 17 (26) | 15 (21)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 16 (22) | 13 (20)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 8 (11)

LIMITATIONS AND CAVEATS:
A DSMB monitored the trial using pre-specified stopping guidelines for efficacy and safety. At the 4th analysis the efficacy bound was crossed. The DSMB determined the study met it's aim and recommended closing the study to enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02054156/SAP_000.pdf
  • Study Protocol (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02054156/Prot_001.pdf